CLINICAL TRIAL: NCT00477802
Title: Botulinum Toxin Type A (Botox) in the Management of Levodopa-Induced Peak-Dose Dyskinesias in Parkinson's Disease: A Double-Blind, Randomized, Placebo Controlled, Cross-Over Design Study
Brief Title: Botulinum Toxin Type A (Botox) in the Management of Levodopa-Induced Peak-Dose Dyskinesias in Parkinson's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Intervention did not appear to be effective in most enrolled patients.
Sponsor: University of Cincinnati (Other)
Collaborators: Allergan (Industry)
Responsible Party: Alberto Espay, MD, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06122801
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; levodopa-induced cervical dyskinesias
MeSH Terms: conditions — Parkinson Disease | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox (Experimental): Randomized into receiving Botox first. At cross-over, patients will receive placebo.
  Interventions: Biological: Botulinum Toxin Type A
- Placebo (Placebo Comparator): Randomized to receive placebo first. At cross-over, patients will receive the active Botox.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Injected once during the course of the study.
  Arms: Botox
Biological: Placebo — Injected once during the course of the study.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether intramuscular injections of botulinum toxin type A (Botox®) in selected cervical muscles at antidystonic dosages can reduce levodopa-induced peak-dose dyskinesias (LID) in the cervical region in adult patients with idiopathic Parkinson's disease. It is hypothesized that the intramuscular injection of antidystonic doses of botulinum toxin into cervical muscles will decrease the duration and severity of LID in the cervical region in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
The study will follow a cross-over design to maximize statistical power and decrease biases inherent to small samples as patients will become their own controls. After a baseline assessment, patients will be randomized to receive either botulinum toxin or an equal amount and distribution of normal saline (placebo). Patients will undergo reassessment of function at one and four weeks after the initial and second session of injections. The second procedure will occur, using the opposite treatment arm (Botox® or saline placebo), three months after the first injection session. Doses of levodopa, dopaminergic agonists, and antidyskinetic drugs if applicable, will be kept constant throughout the study. All study assessments will be carried out at the time treatment is expected to cause the greatest severity of LID.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have idiopathic PD (by standard clinical criteria).
2. Patients must have persistence of LID despite optimization of anti-Parkinsonian medication (duration of LID > 1 [duration of at least 1-25% of the waking time] on item 32 of the United Parkinson's Disease Rating Scale [UPDRS]).
3. Patients must have severity of LID > 1 [mildly disabling] on item 33 of the UPDRS.
4. Patients must have a Mini-Mental State score of > 24.
5. Patients must be willing and able to give consent.

Exclusion Criteria:

1. Patients who are older than 75 years of age.
2. Patients who have a Parkinsonian syndrome that is unresponsive or weakly responsive to levodopa (improvement < 30%).
3. Patients who require concurrent use of warfarin or other anticoagulating agents.
4. Uncontrolled clinically significant medical condition other than the condition under evaluation
5. Known allergy or sensitivity to any of the components in the study medication.
6. Concurrent participation in another investigational drug or device study or participation in the 30 days immediately prior to study enrollment.
7. Any medical condition that may put the subject at an increased risk with exposure to Botox including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function.
8. Evidence of recent alcohol or drug abuse.
9. Infection or skin disorder at an anticipated injection site (if applicable).
10. Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
the change in the "on" time with LID 1 month and 3 months after injected compared to baseline scores. A reduction of 40% in the mean "on" time with LID in the Botox® group compared to the placebo group will be considered significant. | 1 and 3 months after injection

SECONDARY OUTCOMES:
changes in: the duration, severity, and pain of LID using the UPDRS Part IV, physician and patient Clinical Global Impression [CGI] of change, Schwab & England score, Abnormal Involuntary Movement Scale, 4-point modified dyskinesia rating scale (Goetz) | 1 and 3 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Espay, MD, Principal Investigator — University of Cincinnati- Neurology
Locations (1):
- University Neurology - Movement Disorders Clinic, Cincinnati, Ohio, United States